CLINICAL TRIAL: NCT01608464
Title: A Trial Comparing Pre-operative Chemo-radiotherapy With Cisplatin and Fluorouracil Versus Chemotherapy With Docetaxel and Irinotecan in PET Non Responders Resectable Cancer Esophagus: a Multicenter Study
Brief Title: Pre-op Chemo-RT w/CDDP/5FU vs Chemo w/ Docetaxel/Irinotecan in PET Non Responder Resectable Esophagus Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2111-104
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma of Esophagus
Keywords: Randomized trial,; Pre-operative chemo-RT with CDDP and 5-FU; Multicenter study
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Irinotecan; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Arm A: will receive combination of irinotecan and docetaxel regimen for 2 cycles, recycling every 21 days Irinotecan 100 mg/m2 by intra venous infusion over 2 hours in day1 and docetaxel 40 mg/m2 over one hour will be given on day 1 Assessment by PET scan and CT chest and abdomen will be done 2-3 weeks after end of 2nd cycle of irinotecan and docetaxel
  Interventions: Drug: irinotecan and docetaxel
- Arm B (Experimental): Arm B will receive combination of cisplatin, fluorouracil and concurrent radiation therapy 50 Gy in 25 fractions over 5 weeks with cisplatin 75 mg/m2 on first day of week 1 and week 5 and fluorouracil 750 mg/m2 daily by continuous intra venous infusion at Day 1 and Day 29 of Radiation therapy for 4 days.
  PET scan will be repeated 3-4 weeks after end of concurrent chemo-radiation therapy Patients in Arm A and B will go for esophagectomy 4-6 weeks after end of concurrent chemo-radiation therapy or chemotherapy
  Interventions: Drug: Cisplatin, fluorouracil and concurrent radiation therapy

INTERVENTIONS:
Drug: irinotecan and docetaxel — combination of irinotecan and docetaxel regimen for 2 cycles, recycling every 21 days Irinotecan 100 mg/m2 by intra venous infusion over 2 hours in day1 and docetaxel 40 mg/m2 over one hour will be given on day 1 Assessment by PET scan and CT chest and abdomen will be done 2-3 weeks after end of 2nd cycle of irinotecan and docetaxel
  Other Names: Irinotecan; Docetaxel
  Arms: Arm A
Drug: Cisplatin, fluorouracil and concurrent radiation therapy — Cisplatin, fluorouracil and concurrent radiation therapy 50 Gy in 25 fractions over 5 weeks with cisplatin 75 mg/m2 on first day of week 1 and week 5 and fluorouracil 750 mg/m2 daily by continuous intra venous infusion at Day 1 and Day 29 of Radiation therapy for 4 days.
  Other Names: Cisplatin; 5-FU; Concurrent RT with CDDP and 5-FU
  Arms: Arm B

SUMMARY:
The purpose of this study is to improve their outcome by either changing the chemotherapy drugs or giving them radiation therapy with concurrent chemotherapy, hoping that this will improve their outcome.

DETAILED DESCRIPTION:
This study is aimed at improving the outcome of resectable non PET responders, esophageal carcinoma, by either changing the chemotherapy drugs or giving them radiation therapy with concurrent chemotherapy, hoping that this will improve their outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell or adenocarcinoma of the thoracic esophagus and gastro-esophageal junction.
* No distant metastases.
* Signed written informed consent.
* Age less than 75 years.
* Potentially resectable tumor (radiological evidence of resection with no residual disease).
* ECOG 0 to 2.
* Normal serum creatinine and adequate hepatic function, serum bilirubin less than 30 mmol/l, serum alkaline phosphatase less than 2 times upper limit of normal and ALT and AST of less than 4 upper limits of normal.
* Normal bone marrow function with absolute neutrophile count of more than 1500/ml, hemoglobin more than 80 gm/L and platelets more than 100,000 /ml

Exclusion Criteria:

1. Serious underlying medical condition which could impair the patient ability to participate in the clinical trial or comply to follow up
2. Prior treatment with other anti cancer therapy or radiation therapy.
3. Legal incapacity.
4. Previous malignancy within 5 years except adequately treated non melanomatous skin cancer or in situ cervical cancer.
5. Psychiatric or mental disorder precluding the understanding of the information of the trial topics and giving valid informed consent.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response ( regression score 1a- see response assessment) in each treatment group | 5 yrs

SECONDARY OUTCOMES:
Rate of conversion from PET non responder to responder with each type of salvage therapy | 5 yrs
  * Failure Free Survival for each treatment group
  * Overall Survival for each treatment group
  * ERCC1 as a predictor of failure of response to cisplatin based chemotherapy in neo adjuvant setting.

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided